CLINICAL TRIAL: NCT06938451
Title: A Real-world Study of FGF19 Overexpression Status and Treatment Outcome and Prognosis in Advanced Hepatocellular Carcinoma
Brief Title: Relationship Between FGF19 Overexpression and Disease Prognosis
Acronym: FGF19
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, ZHAO YING, Principal Investigator, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: V1.0 20250309
Record Dates: First submitted 2025-03-27; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: FGF19; hepatocellular carcinoma; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- inspection team: Surgically resected liver tissue samples were sent to a third-party pathology slice reviewer for uniform reading, and a report on FGF19 expression results was issued and returned to the project team. The clinical data of the patient will be collected at the same time.

INTERVENTIONS:
Other:  — This is an observational study and does not involve an intervention

SUMMARY:
A real-world study of FGF19 overexpression status and treatment outcome and prognosis in advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
This is a real-world, single-arm, observational study to collect information on the diagnosis and prognosis of hepatocellular carcinoma patients with previous tissue samples in routine clinical practice, and to detect the expression of FGF19 expression in tissue samples, with a view to discovering prognostic and predictive markers for advanced hepatocellular carcinoma The treatment protocol of this study follows the clinical practice and does not set any limitations on the interventions for patients.

In this study, real-world liver tissue samples will be collected from patients with hepatocellular liver cancer after surgical resection, and the samples will be sent to a third-party pathology slice reviewer for review, and a report on the FGF19 expression results will be returned to the project team. Simultaneously collect clinical data of the patient.

According to the principle of clinical routine diagnosis and treatment, the patient's imaging data were collected, and the imaging of the 2-month period was evaluated, and whether the disease progressed was judged according to the RESCIST v1.1 standard. Every two months will be an observation cycle. Each subject will be followed from the first treatment until disease progression or change of drug regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years on the day of signing the informed consent form
* Histologically or clinically confirmed diagnosis of intermediate to advanced HCC
* Adequate tissue samples of previous liver cancer
* Expected survival of more than 3 months

Exclusion Criteria:

* Fibrous laminae or sarcomatoid HCC or mixed HCC-ICC, or other rare non-HCC pathologic subtypes
* Other conditions that, in the opinion of the investigator, make participation in this trial inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC in the middle to late stages of the disease；Sufficient previous hepatocellular carcinoma tissue samples were available for immunohistochemical detection of FGF19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Enrollment until disease progression
  PFS was calculated from the date of randomization to the date of the first documented disease progression, with no time constraints involved, marked by the appearance of disease progression
OS | Start of enrollment until death (from any cause)
  Observation until death from the beginning of participation in the study observation until death from any cause, no time frame limitations were involved. Calculation of OS based on time of death

SECONDARY OUTCOMES:
ORR | Time to enrollment until disease downsizing
  Proportion of patients whose tumor volume shrinks to a preset value and remains unchanged for a given period of time, total study duration 36 months, ORR observation period within 36 months

CONTACTS AND LOCATIONS:
Overall Officials: ZHAOYING Resident physician, phD, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided